CLINICAL TRIAL: NCT02196532
Title: Retinal Nerve Fiber Layer Thickness Changes in Migraine: A Meta-Analysis of Case-control Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yifan Feng (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor-Investigator, Yifan Feng, Zhongshan hospital, Fudan University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: FYF20140717
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Migraine
Keywords: retinal nerve fiber layer thickness; optical coherence tomography; migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- migraine group: Patients with migraine
  Interventions: Device: Device: Optical coherence tomography
- healthy control: Sex- and agematched healthy subjects
  Interventions: Device: Device: Optical coherence tomography

INTERVENTIONS:
Device: Device: Optical coherence tomography

SUMMARY:
Optical coherence tomography (OCT) is a non-invasive retinal imaging technology that can provide high-resolution cross-sectional images of the peripapillary retinal nerve fiber layer (RNFL) and measure its thickness. A reduction of the RNFL thickness has been detected in several neurodegenerative diseases, such as multiple sclerosis, CADASIL and Alzheimer's disease. Different studies have reported RNFL changes also in migraine, is a common hereditary chronic neurovascular disorder, characterized by dysfunction of the autonomic nervous system. The pathophysiology of migraine has not been fully clarified, but there is increasing evidence that episodes of migraine with aura are initiated by a focal reduction in cerebral blood flow, which occurs most commonly in the posterior region of one hemisphere. Although vasoconstriction of cerebral and retinal blood vessels is a transient phenomenon, the chronic nature of the migraine might cause permanent structural abnormalities of the brain and also of the retina, which may correlate with RNFL thinning. Previous studies on this subject, however, reported contradicting results. Some investigations reported reductions of the RNFL thickness while others did not. In the present study, in order to determine whether RNFL thickness is reduced in migraine patients, the investigators performed a meta-analysis and systematically evaluated RNFL thickness measurements with OCT in a series of migraine patients and in the healthy control groups.

ELIGIBILITY:
Inclusion Criteria:

1. case-control studies;
2. patients with Migraine were compared with healthy controls;
3. all subjects underwent RNFL thickness measurement by OCT;
4. studies should provide the data of peripapillary RNFL thickness;
5. sample size ≥10 in each group.

Exclusion Criteria:

1. authors did not make RNFL measurements;
2. study without healthy control group;
3. the outcome values can not be used for meta-analysis;
4. duplicated articles.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migraine patients and healthy subjects were included and underwent OCT examinations
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer Thickness | Baseline
  Retinal nerve fiber layer thickness included average thickness (360° measurement), temporal quadrant thickness (316-45°), superior quadrant thickness (46-135°), nasal quadrant thickness (136-225°) and inferior quadrant thickness (226-315°)was measured by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Feng, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China